CLINICAL TRIAL: NCT02552823
Title: A Randomized, Controlled, Cross-over Trial Examining the Effect of Peas on Post-prandial Glucose Response in Healthy Adults
Brief Title: Effects of Peas on Blood Glucose Control
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: St. Boniface Hospital (Other)
Collaborators: Agriculture and Agri-Food Canada (Other Government)
Responsible Party: Principal Investigator, Dr. Heather Blewett, Principal Investigator, St. Boniface Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: H29
Record Dates: First submitted 2015-07-27; First posted 2015-09-17 (Estimated); Last update posted 2024-02-02 (Actual); Status verified 2024-01

CONDITIONS: Post-prandial Glucose Response

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (10):
- White bread 1 (Placebo Comparator): Groups 1 and 2, Visit 1 White bread (equal to 50g available carbohydrate) given to fasting participant
  Interventions: Other: Group1; Other: Group2
- Pea variety 1 with rice (Experimental): Group 1,Visit 2-5 Pea variety 1 with rice (25g available carbohydrate of each) given as breakfast to fasting participants
  Interventions: Other: Group1
- Pea variety 2 with rice (Experimental): Group 1, Visit 2-5 Pea variety 2 with rice (25g available carbohydrate of each) given as breakfast to fasting participants
  Interventions: Other: Group1
- Pea variety 3 with rice (Experimental): Group 1, Visit 2-5 Pea variety 3 with rice (25g available carbohydrate of each) given as breakfast to fasting participants
  Interventions: Other: Group1
- Rice (Experimental): Group 1, Visit 2-5 Rice (equal to 50g available carbohydrate) given as breakfast to fasting participants
  Interventions: Other: Group1
- White bread 2 (Placebo Comparator): Groups 1 and 2, Visit 6 White bread (equal to 50g available carbohydrate) given to fasting participant
  Interventions: Other: Group1; Other: Group2
- Pea variety 1 with potato (Experimental): Group 2, Visit 2-5 Pea variety 1 with potato (25g available carbohydrate of each) given as breakfast to fasting participants
  Interventions: Other: Group2
- Pea variety 2 with potato (Experimental): Group 2, Visit 2-5 Pea variety 2 with potato (25g available carbohydrate of each) given as breakfast to fasting participants
  Interventions: Other: Group2
- Pea variety 3 with potato (Experimental): Group 2, Visit 2-5 Pea variety 3 with potato (25g available carbohydrate of each) given as breakfast to fasting participants
  Interventions: Other: Group2
- Potato (Experimental): Group2, Visit 2-5 Potato (equal to 50g available carbohydrate) given as breakfast to fasting participants
  Interventions: Other: Group2

INTERVENTIONS:
Other: Group1
  Other Names: Peas with Rice
  Arms: Pea variety 1 with rice; Pea variety 2 with rice; Pea variety 3 with rice; Rice; White bread 1; White bread 2
Other: Group2
  Other Names: Peas with potato
  Arms: Pea variety 1 with potato; Pea variety 2 with potato; Pea variety 3 with potato; Potato; White bread 1; White bread 2

SUMMARY:
Diabetes is one of the most common chronic diseases affecting Canadians (PHAC, 2011). Lifestyle modifications that include a diet high in fibre may lower the risk of developing type 2 diabetes (CDA, 2013). In this context, the presence of fibre in carbohydrate rich foods has been widely recognized for its effect on post-prandial glucose response (PPGR). Peas are high in fibre and protein and show great potential as a functional food. A health claim for PPGR would increase market demand for peas, and help those who want to limit the rise in blood sugar after a meal choose products to meet their goals, but there are several gaps in the literature that need to be filled before a submission to Health Canada can be successful: 1) test foods in appropriate serving sizes; 2) test both the glucose and insulin response; 3) test varieties of peas that that currently available on the market; 4) test whole/split peas (not fractions or isolates); 5) compare peas to appropriate starchy reference food (rice or potato). The proposed study design will address all of these gaps in the current literature and take into consideration Health Canada's guidance document for health claims related to the reduction in PPGR, which sets out the criteria by which the validity of such claims will be assessed.

Specific objectives

1. To determine the effect of 3 common market classes of peas on PPGR and insulin response in a cross-over, randomized, controlled clinical trial.
2. To assess the effect of 3 common market classes of peas on appetite-related sensations using visual analog scales.
3. To demonstrate whether the test and reference products were liked or disliked similarly by participants.
4. To assess any gastrointestinal side effects from eating the test products

DETAILED DESCRIPTION:
A randomized, controlled, cross-over study designed to examine the PPGR to peas will be conducted at the I.H. Asper Clinical Research Institute in Winnipeg, Manitoba. The study will be divided into 2 groups of 24 healthy volunteers each. In Group 1, eligible participants who have provided consent will be asked to attend 6 clinic visits in a fasted state. Participants will be given white bread at their first and last visits, peas with rice at 3 visits and rice at 1 visit. At each visit participants will provide 7 blood samples via finger poke, 6 questionnaires about their appetite and a questionnaire about the acceptability of the test food. Each visit will last approximately 2.5h and be separated by 3-10 days. Group 2 will undergo the exact same study procedures as group 1, but rice will be replaced with potato.

ELIGIBILITY:
Inclusion criteria

1. Generally healthy male or female, between the age of 18-40 years;
2. Body mass index (BMI) 18.5-34.5 kg/m2;
3. HbA1c <6.0%;
4. Willing to provide informed consent;
5. Willing/able to comply with the requirements of the study.

Exclusion criteria

1. Pregnant or lactating;
2. Medical history of diabetes mellitus, fasting plasma glucose ≥7.0 mmol/L or use of insulin or oral medication to control blood sugar;
3. Medical history of cardiovascular disease
4. Systolic blood pressure >140 mmHg or diastolic blood pressure >90 mmHg;
5. Fasting plasma total cholesterol >7.8 mmol/L;
6. Fasting plasma HDL <0.9 mmol/L;
7. Fasting plasma LDL >5.0 mmol/L;
8. Fasting plasma triglycerides >2.3 mmol/L;
9. A change in blood glucose concentration less than 1 mmol/L between baseline and 30 minutes after consumption of white bread at visit 1;
10. Maximum blood glucose concentration occurs after 60 minutes after consumption of white bread at visit 1;
11. Major surgery within the last 3 months;
12. Medical history of inflammatory disease (ie. Systemic lupus erythematosis, rheumatoid arthritis, psoriasis) or use of any corticosteroid medications within 3 months;
13. Medical history of liver disease or liver dysfunction (defined as plasma AST or ALT ≥1.5 times the upper limit of normal (ULN));
14. Medical history of kidney disease or kidney dysfunction (defined as blood urea nitrogen and creatinine ≥ 1.8 times the ULN));
15. Presence of a gastrointestinal disorder, daily use of any stomach acid-lowering medications or laxatives (including fibre supplements) within the past month or antibiotic use with the past 6 weeks;
16. Active treatment for any type of cancer within 1 year prior to study start;
17. Other medical, psychiatric, or behavioral factors that in the judgment of the principal Investigator may interfere with study participation or the ability to follow the intervention protocol;
18. Shift worker;
19. Tobacco use current or within the last 3 months;
20. Allergies to peas;
21. Aversion or unwillingness to eat study foods;
22. Consuming >4 servings of pulses per week;
23. Use of any prescription or non-prescription drug, herbal or nutritional supplement known to affect glycemia;
24. Participation in another clinical trial, current or in the past 4 weeks;
25. Unstable body weight (defined as >5% change in 3 months) or actively participating in a weight loss program.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2015-10-16 (Actual); Primary Completion 2017-08-14 (Actual); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Postprandial blood glucose | up to 2 hours following a meal
  samples collected to test glucose at fasting and at 15,30,45,60,90 and 120 minutes after the first bite of the test product
Postprandial blood insulin | up to 2 hours following a meal
  samples collected to test insulin at fasting and at 15,30,45,60,90 and 120 minutes after the first bite of the test product

SECONDARY OUTCOMES:
Hunger (Visual analogue scales) | up to 2 hours following a meal
  Visual analogue scales are administered pre-meal, immediately post-meal and 30, 60, 90 and 120 minutes
Fullness (Visual analogue scales) | up to 2 hours following a meal
  Visual analogue scales are administered pre-meal, immediately post-meal and 30, 60, 90 and 120 minutes
Desire to eat (Visual analogue scales) | up to 2 hours following a meal
  Visual analogue scales are administered pre-meal, immediately post-meal and 30, 60, 90 and 120 minutes

OTHER OUTCOMES:
Acceptability of test products based on sensory scales | immediately after eating test product
  scales will assess overall, colour, aroma, flavour and texture likeability
Gastrointestinal side effects | up to 24 hours following a meal
  After consumption of the test product, any abnormal gastrointestinal side effects will be recorded

CONTACTS AND LOCATIONS:
Overall Officials: Heather J Blewett, PhD, Principal Investigator — Agriculture and Agri-Food Canada
Locations (1):
- I. H. Asper Clinical Research Institute, Winnipeg, Manitoba, Canada

REFERENCES:
- [Background] Hamberg O, Rumessen JJ, Gudmand-Hoyer E. Blood glucose response to pea fiber: comparisons with sugar beet fiber and wheat bran. Am J Clin Nutr. 1989 Aug;50(2):324-8. doi: 10.1093/ajcn/50.2.324. PMID 2547300
- [Background] Marinangeli CP, Jones PJ. Chronic intake of fractionated yellow pea flour reduces postprandial energy expenditure and carbohydrate oxidation. J Med Food. 2011 Dec;14(12):1654-62. doi: 10.1089/jmf.2010.0255. PMID 22145774
- [Background] Marinangeli CP, Kassis AN, Jones PJ. Glycemic responses and sensory characteristics of whole yellow pea flour added to novel functional foods. J Food Sci. 2009 Nov-Dec;74(9):S385-9. doi: 10.1111/j.1750-3841.2009.01347.x. PMID 20492127
- [Background] Mollard RC, Wong CL, Luhovyy BL, Cho F, Anderson GH. Second-meal effects of pulses on blood glucose and subjective appetite following a standardized meal 2 h later. Appl Physiol Nutr Metab. 2014 Jul;39(7):849-51. doi: 10.1139/apnm-2013-0523. Epub 2014 May 5. PMID 24797207
- [Background] Mollard RC, Zykus A, Luhovyy BL, Nunez MF, Wong CL, Anderson GH. The acute effects of a pulse-containing meal on glycaemic responses and measures of satiety and satiation within and at a later meal. Br J Nutr. 2012 Aug;108(3):509-17. doi: 10.1017/S0007114511005836. Epub 2011 Nov 7. PMID 22054112
- [Background] Mollard RC, Wong CL, Luhovyy BL, Anderson GH. First and second meal effects of pulses on blood glucose, appetite, and food intake at a later meal. Appl Physiol Nutr Metab. 2011 Oct;36(5):634-42. doi: 10.1139/h11-071. Epub 2011 Sep 29. PMID 21957874
- [Background] Schafer G, Schenk U, Ritzel U, Ramadori G, Leonhardt U. Comparison of the effects of dried peas with those of potatoes in mixed meals on postprandial glucose and insulin concentrations in patients with type 2 diabetes. Am J Clin Nutr. 2003 Jul;78(1):99-103. doi: 10.1093/ajcn/78.1.99. PMID 12816777
- [Background] Sievenpiper JL, Kendall CW, Esfahani A, Wong JM, Carleton AJ, Jiang HY, Bazinet RP, Vidgen E, Jenkins DJ. Effect of non-oil-seed pulses on glycaemic control: a systematic review and meta-analysis of randomised controlled experimental trials in people with and without diabetes. Diabetologia. 2009 Aug;52(8):1479-95. doi: 10.1007/s00125-009-1395-7. Epub 2009 Jun 13. PMID 19526214